CLINICAL TRIAL: NCT03548467
Title: An Open Labelled First Human Dose Phase 1/2a Study to Evaluate Safety, Feasibility, Efficacy of Multiple Dosing With Individualised VB10.NEO and Bempegaldesleukin (NKTR-214) Immunotherapy in Patients With Locally Advanced or Metastatic Melanoma, Non-small Cell Lung Cancer (NSCLC), Clear Renal Cell Carcinoma, Urothelial Cancer or Squamous Cell Carcinoma of Head and Neck, Who Did Not Reach Complete Responses With Current Standard of Care Immune Checkpoint Blockade
Brief Title: A Study to Evaluate Safety and Efficacy of Multiple Dosing With VB10.NEO and Bempegaldesleukin (NKTR-214) Immunotherapy in Patients With Locally Advanced or Metastatic Cancer
Acronym: DIRECT-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nykode Therapeutics ASA (Industry)
Collaborators: Nektar Therapeutics (Industry); Vaccibody AS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB N-01
Record Dates: First submitted 2018-04-17; First posted 2018-06-07 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced or Metastatic Solid Tumours
Keywords: melanoma; NSCLC; clear renal cell carcinoma; urothelial cancer or SCCHN
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell | interventions — bempegaldesleukin

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VB10.NEO intervention (Experimental): Treatment with individualized VB10.NEO immunotherapy will commence as soon as the patient-specific VB10.NEO vaccine is available and if the patient-specific vaccine meets all pre-specified product release criteria after manufacturing to patients within the selected tumor types.
  Interventions: Biological: VB10.NEO
- VB10.NEO in combination with bempegaldesleukin (NKTR-214) (Experimental): Bempegaldesleukin (NKTR-214) will be given in combination with VB10.NEO in up to 10 patients with SCCHN. Treatment with individualized VB10.NEO immunotherapy will commence as soon as the patient-specific VB10.NEO vaccine is available and if the patient-specific vaccine meets all pre-specified product release criteria after manufacturing. Bempegaldesleukin (NKTR-214) will be given after at least 4 doses of VB10.NEO.
  Interventions: Biological: VB10.NEO; Drug: Bempegaldesleukin

INTERVENTIONS:
Biological: VB10.NEO — VB10.NEO is a vaccine and is supplied as a sterile, ready to use solution (14 vaccinations will be given).
Drug: Bempegaldesleukin — 0.006 mg/kg bempegaldesleukin (NKTR-214) will be administered intravenously q4w for up to 11 doses starting from week 11 or at any dosing visit up to week 34 and for up to week 50 (up to 11 doses). The first 2 doses will be in a Q3W interval and following doses in Q4W intervals.
  Other Names: NKTR-214
  Arms: VB10.NEO in combination with bempegaldesleukin (NKTR-214)

SUMMARY:
This open labelled first in human dose phase 1/2a study is designed to evaluate safety, feasibility and efficacy of multiple dosing with individualised VB10.NEO and bempegaldesleukin (NKTR-214) immunotherapy in patients with locally advanced or metastatic solid tumours.

DETAILED DESCRIPTION:
This open labelled first in human dose phase 1/2a study is designed to evaluate safety, feasibility and efficacy of multiple dosing with individualised VB10.NEO immunotherapy in patients with locally advanced or metastatic solid tumours including melanoma, non-small cell lung cancer (NSCLC), clear renal cell carcinoma, urothelial cancer or squamous cell carcinoma of the head and neck (SCCHN), who did not reach complete responses with immune checkpoint inhibitor (CPI) therapy as their standard of care (SOC) treatment.

Patients with melanoma, NSCLC, RCC and urothelial carcinoma must upon screening, have been receiving a CPI (anti-PD-1 or anti-PD-L1) for at least 12 weeks as the patient's standard of care. Patients with SCCHN can be screened as long as they have initiated treatment with CPI as SOC. The VB10.NEO vaccine will be added to continuing CPI treatment and shall not replace, omit, postpone or terminate the standard therapy. Patients who have been treated with CPI for at least 12 weeks, will be enrolled in case of some benefit to CPI treatment is expected, as defined by partial response, stable disease or disease progression (in case of a mixed response to CPI, provided at least one lesion shows measurable regression and patient, according to the investigator, would have a clinical benefit of continued immunotherapy).

The assumption is to combine the immuno-stimulating effect of CPIs with immune responses towards specific neo-antigens in the vaccine, which may possibly increase the anti-tumour effect to reach durable efficacy.

One arm of the study patients with SCCHN will have the option to be treated with bempegaldesleukin (NKTR-214) in combination with personalised VB10.NEO. This arm is open for enrollment from November 2019.

The study will be conducted in two parts. Part A will evaluate safety, feasibility and efficacy of individualised VB10.NEO and bempegaldesleukin (NKTR-214) immunotherapy in SCCHN patients. The expansion part B will explore efficacy and safety in further patients with selected types of cancer showing signs of efficacy during part A.

ELIGIBILITY:
Inclusion criteria for all arms

* Have histologically confirmed locally advanced or metastatic melanoma, NSCLC, RCC, urothelial carcinoma or SCCHN.
* Patients must have been on CPI (i.e., anti-PD-1 or anti PD-L1) for at least 12 weeks before screening and must be on CPI treatment as part of their cancer treatment as prescribed by the treating physician.

Inclusion criteria for SCCHN only

• Patients must be on CPI or must initiate treatment with CPI at screening as part of their cancer treatment.

All arms

* Patients who have been on CPI for longer than 12 weeks at screening need to be per RECIST:

  * in partial response or;
  * stable disease or,
  * in progression, i.e., in case of a mixed response to CPI, provided at least one lesion shows measurable regression and who, according to the investigator, have a clinical benefit of continued immunotherapy.
* Adequate tumour specimen must be available for exome sequencing.
* Measurable disease per RECIST 1.1 criteria.
* ECOG performance status ≤ 1.
* Life expectancy at least 6 months in the best judgement of the investigator.
* Willing and able to sign a written informed consent form.

Exclusion criteria

* Ocular melanoma.
* Brain metastases (unless controlled and stable for at least 6 weeks) or leptomeningeal spread of disease.
* Positive serological test for hepatitis C virus or hepatitis B virus surface antigen (HBsAg) or human immunodeficiency virus (HIV).
* Other concomitant or prior malignant disease, except for adequately treated basal cell carcinoma or other non-melanomatous skin cancer, low-grade urothelial cancer or other malignancies treated with curative intent within 2 or more years pre-study entry and in complete remission at study entry
* Patients who have an active, known or suspected autoimmune disease. Patients having required systemic treatment within the past 3 months or have a documented history of clinically severe autoimmune disease that require systemic steroids or immunosuppressive agents (Exceptions include any patient on 10 mg or less of prednisolone or equivalent, patients with vitiligo, hypothyroidism stable on hormone replacement; type 1 diabetes, Grave's disease, Hashimoto's disease, alopecia areata, eczema).
* Immunosuppression including the continued use (> 7 days) of high-dose (>10 mg of prednisolone or equivalents) systemic steroids or the use of immunosuppressive agents for any concurrent condition.

Other protocol defined inclusion exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of Adverse Events including SAEs (Safety/tolerability) of VB10.NEO and the combination of VB10.NEO and bempegaldesleukin (NKTR-214) | Up to 24 months
  Total number, severity (CTCAE grade) of adverse events (AEs), and if AE is leading to treatment discontinuation.

SECONDARY OUTCOMES:
Immunogenicity by T-cell activity to each neoepitope of VB10.NEO and the combination of VB10.NEO and bempegaldesleukin (NKTR-214) | Up to 24 months
  Descriptive analyses for each patient of the immune-response to each neoepiotope
Objective Response Rate (ORR) | Up to 24 months
  Description of tumor response by iRECIST at regular intervals
Duration of Response (DOR) | Up to 24 months
  Descriptive analysis of DOR by iRECIST at regular intervals
Progression-free survival (PFS) | Up to 24 months
  Descriptive analysis of PFS by iRECIST at regular intervals
Survival at end of treatment (EoT) and end of study (EoS) | At 14 months and 24 months
  Proportion of patients who are alive at EoT and EoS

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Charité Research Organisation, Campus Benjamin Franklin, Berlin
  - Krankenhaus Nordwest gGmbH, Frankfurt
  - Martin-Luther-Universität Halle-Wittenberg, Universitätsklinikum Halle (Saale), Halle
  - University Hospital Heidelberg, NCT, Im Neuenheimer Feld 460, Heidelberg
  - Universitätsmedizin Mannheim, Mannheim
  - Klinik und Poliklinik für Innere Medizin III, Hämatologie und Onkologie, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srikrishna D, Sachsenmeier K. We need to bring R0 < 1 to treat cancer too. Genome Med. 2021 Jul 26;13(1):120. doi: 10.1186/s13073-021-00940-9. PMID 34311780